CLINICAL TRIAL: NCT02870101
Title: Performance of Nucleic Acid Amplification Tests for the Detection of Neisseria Gonorrhoeae and Chlamydia Trachomatis in Extragenital Sites
Brief Title: Performance of Nucleic Acid Amplification Tests for the Detection of NG and CT
Acronym: pNAAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00073558; 5UM1AI104681 (NIH)
Record Dates: First submitted 2016-08-12; First posted 2016-08-17 (Estimated); Results first posted 2019-04-26 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Neisseria Gonorrhoeae Infection; Chlamydia Trachomatis Infection; Sexually Transmitted Infections
Keywords: Nucleic acid amplification tests; Neisseria gonorrhoeae infection; Chlamydia trachomatis infection; Sexually transmitted infection; Pharynx; Rectum; Gram-Negative Bacterial Infections; Bacterial Infections; Genital Diseases, Male; Genital Diseases, Female
MeSH Terms: conditions — Gonorrhea; Sexually Transmitted Diseases; Gram-Negative Bacterial Infections; Bacterial Infections; Genital Diseases, Male; Genital Diseases, Female

STUDY DESIGN:
Masking Description: All information collected anonymously.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention (Other): Performance of three nucleic acid amplification tests (NAATs) to detect Neisseria gonorrhoeae (NG) and Chlamydia trachomatis (CT) from swabs collected from the pharynx and rectum. Assays include: Nucleic acid amplification test 1 for NG and CT; Nucleic acid amplification test 2 for NG and CT; and, Nucleic acid amplification test 3 for NG and CT.
  Interventions: Diagnostic Test: Nucleic acid amplification test 1 for NG and CT; Diagnostic Test: Nucleic acid amplification test 2 for NG and CT; Diagnostic Test: Nucleic acid amplification test 3 for NG and CT

INTERVENTIONS:
Diagnostic Test: Nucleic acid amplification test 1 for NG and CT — A combination test using real-time PCR to detect DNA from NG and CT.
Diagnostic Test: Nucleic acid amplification test 2 for NG and CT — A combination test using target amplification to detect RNA from NG and CT.
Diagnostic Test: Nucleic acid amplification test 3 for NG and CT — A combination test using real-time PCR to detect DNA from NG and CT.

SUMMARY:
The purpose of this study was to use participant samples to simultaneously evaluate three nucleic acid amplification tests (NAATs) diagnostic platforms.

DETAILED DESCRIPTION:
Background & Significance: Infections due to Neisseria gonorrhoeae (NG) and Chlamydia trachomatis (CT) are major threats to public health. Most CT and NG infections are asymptomatic, but infection can lead to serious sequelae, including infertility, chronic pelvic pain, adverse obstetrical outcomes, increased risk of acquiring the human immunodeficiency virus (HIV), and disseminated infection.

There has also been growing concern over antibiotic resistance. In 2013, the US Centers for Disease Control and Prevention (CDC) classified drug-resistant NG as one of the three urgent-level resistant bacteria. Improved detection of extragenital NG is thought to be a crucial component of adequate treatment and for prevention of further resistance.

Currently, the CDC recommends using NAATs to screen and diagnose for NG and CT in the genitourinary tract due to their superior sensitivity compared to traditional culture methods. There are currently no FDA-approved commercial NAAT tests for the detection of pharyngeal and rectal NG or CT infections. The goal of this study is to evaluate the diagnostic performance of three NAAT assays for detection of extragenital NG and CT infections.

Design & Procedures: A cross-sectional, single visit study evaluating the performance of three commercial NAATs to detect NG and CT in the rectum and pharynx. A fourth NAAT will be used as a tiebreaker. The performance of the fourth NAAT will not be evaluated. Each manufacturer will provide a specific swab collection kit and transport media.

This research study will take place at healthcare clinics that focus on sexually transmitted infections, women's health, student health, family planning, and lesbian, gay, bisexual, and transgender (LGBT) health. This research will include specimens collected from adult males, females, and transgender persons seeking sexually transmitted infection (STI) testing at the participating study clinics. Both symptomatic and asymptomatic participants are included in the study population.

Potential participants will be identified, assessed for eligibility, and asked to provide oral informed consent. If a potential participant agrees to take part in the research, the participant will have eight total swabs collected: four swabs from the pharynx and four swabs from the rectum. The swabs needed for routine clinical care are taken first prior to collection of the research study swabs. All study procedures take place during one clinic visit; there are no follow-up visits as part of the study. Participants continue with routine clinical care as directed by their medical providers.

Subject participation is confidential and anonymous. The results of the tests and participation in this research are not placed in the participant's medical records.

Each study swab is used for a specific NAAT and tested at one of the two reference testing laboratories. The Anatomic Site Infection Status (ASIS) is defined by the results of the two other NAATs, and, if necessary, results from the tiebreaker NAAT. Each anatomic site is considered in isolation. If fewer than four swabs at an anatomic site are completed, then the test results from that specific anatomic site are excluded from analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Attending a participating clinic for evaluation of sexually transmitted infections (STIs)
2. ≥18 years of age at date of screening
3. Able and willing to provide informed consent
4. Willing to comply with study procedures, including collection of 4 swabs each from the pharynx and rectum for NG and CT testing

Exclusion Criteria:

1. Receipt of any systemic antibacterial drug in the past 14 days
2. Receipt of myelosuppressive chemotherapy in the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2767 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D Klausner, MD, MPH, Principal Investigator — UCLA David Geffen School of Medicine and Fielding School of Public Health
Locations (9):
- United States (9):
  - AIDS Health Foundation - Hollywood, Hollywood, California
  - Los Angeles LGBT Clinic, Los Angeles, California
  - Denver Health and Hospital Authority, Denver, Colorado
  - AIDS Healthcare Foundation - Miami, Miami, Florida
  - University of Miami, Miami, Florida
  - Louisiana State University, New Orleans, Louisiana
  - Wayne State University, Detroit, Michigan
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Central Texas Clinical Research, Austin, Texas

REFERENCES:
- [Background] Liu B, Roberts CL, Clarke M, Jorm L, Hunt J, Ward J. Chlamydia and gonorrhoea infections and the risk of adverse obstetric outcomes: a retrospective cohort study. Sex Transm Infect. 2013 Dec;89(8):672-8. doi: 10.1136/sextrans-2013-051118. Epub 2013 Sep 4. PMID 24005255
- [Background] O'Brien JP, Goldenberg DL, Rice PA. Disseminated gonococcal infection: a prospective analysis of 49 patients and a review of pathophysiology and immune mechanisms. Medicine (Baltimore). 1983 Nov;62(6):395-406. PMID 6415361
- [Background] Westrom L, Joesoef R, Reynolds G, Hagdu A, Thompson SE. Pelvic inflammatory disease and fertility. A cohort study of 1,844 women with laparoscopically verified disease and 657 control women with normal laparoscopic results. Sex Transm Dis. 1992 Jul-Aug;19(4):185-92. PMID 1411832
- [Background] Rottingen JA, Cameron DW, Garnett GP. A systematic review of the epidemiologic interactions between classic sexually transmitted diseases and HIV: how much really is known? Sex Transm Dis. 2001 Oct;28(10):579-97. doi: 10.1097/00007435-200110000-00005. PMID 11689757
- [Background] Deguchi T, Yasuda M, Ito S. Management of pharyngeal gonorrhea is crucial to prevent the emergence and spread of antibiotic-resistant Neisseria gonorrhoeae. Antimicrob Agents Chemother. 2012 Jul;56(7):4039-40; author re[ply 4041-2. doi: 10.1128/AAC.00505-12. No abstract available. PMID 22700700
- [Background] Workowski KA, Bolan GA; Centers for Disease Control and Prevention. Sexually transmitted diseases treatment guidelines, 2015. MMWR Recomm Rep. 2015 Jun 5;64(RR-03):1-137. PMID 26042815
- [Background] Zakher B, Cantor AG, Pappas M, Daeges M, Nelson HD. Screening for gonorrhea and Chlamydia: a systematic review for the U.S. Preventive Services Task Force. Ann Intern Med. 2014 Dec 16;161(12):884-93. doi: 10.7326/M14-1022. PMID 25244000
- [Background] Ota KV, Tamari IE, Smieja M, Jamieson F, Jones KE, Towns L, Juzkiw J, Richardson SE. Detection of Neisseria gonorrhoeae and Chlamydia trachomatis in pharyngeal and rectal specimens using the BD Probetec ET system, the Gen-Probe Aptima Combo 2 assay and culture. Sex Transm Infect. 2009 Jun;85(3):182-6. doi: 10.1136/sti.2008.034140. Epub 2009 Jan 6. PMID 19126571
- [Background] Schachter J, Moncada J, Liska S, Shayevich C, Klausner JD. Nucleic acid amplification tests in the diagnosis of chlamydial and gonococcal infections of the oropharynx and rectum in men who have sex with men. Sex Transm Dis. 2008 Jul;35(7):637-42. doi: 10.1097/OLQ.0b013e31817bdd7e. PMID 18520976
- [Background] Trebach JD, Chaulk CP, Page KR, Tuddenham S, Ghanem KG. Neisseria gonorrhoeae and Chlamydia trachomatis among women reporting extragenital exposures. Sex Transm Dis. 2015 May;42(5):233-9. doi: 10.1097/OLQ.0000000000000248. PMID 25868133
- [Background] Bachmann LH, Johnson RE, Cheng H, Markowitz L, Papp JR, Palella FJ Jr, Hook EW 3rd. Nucleic acid amplification tests for diagnosis of Neisseria gonorrhoeae and Chlamydia trachomatis rectal infections. J Clin Microbiol. 2010 May;48(5):1827-32. doi: 10.1128/JCM.02398-09. Epub 2010 Mar 24. PMID 20335410
- [Background] Cosentino LA, Campbell T, Jett A, Macio I, Zamborsky T, Cranston RD, Hillier SL. Use of nucleic acid amplification testing for diagnosis of anorectal sexually transmitted infections. J Clin Microbiol. 2012 Jun;50(6):2005-8. doi: 10.1128/JCM.00185-12. Epub 2012 Apr 4. PMID 22493338
- [Background] Geelen TH, Rossen JW, Beerens AM, Poort L, Morre SA, Ritmeester WS, van Kruchten HE, van de Pas MM, Savelkoul PH. Performance of cobas(R) 4800 and m2000 real-time assays for detection of Chlamydia trachomatis and Neisseria gonorrhoeae in rectal and self-collected vaginal specimen. Diagn Microbiol Infect Dis. 2013 Oct;77(2):101-5. doi: 10.1016/j.diagmicrobio.2013.06.020. Epub 2013 Jul 23. PMID 23891224
- [Background] Moncada J, Schachter J, Liska S, Shayevich C, Klausner JD. Evaluation of self-collected glans and rectal swabs from men who have sex with men for detection of Chlamydia trachomatis and Neisseria gonorrhoeae by use of nucleic acid amplification tests. J Clin Microbiol. 2009 Jun;47(6):1657-62. doi: 10.1128/JCM.02269-08. Epub 2009 Apr 15. PMID 19369445
- [Background] Perry MD, Jones RN, Corden SA. Is confirmatory testing of Roche cobas 4800 CT/NG test Neisseria gonorrhoeae positive samples required? Comparison of the Roche cobas 4800 CT/NG test with an opa/pap duplex assay for the detection of N gonorrhoeae. Sex Transm Infect. 2014 Jun;90(4):303-8. doi: 10.1136/sextrans-2013-051410. Epub 2014 Mar 20. PMID 24653040
- [Background] Harryman L, Scofield S, Macleod J, Carrington D, Williams OM, Fernandes A, Horner P. Comparative performance of culture using swabs transported in Amies medium and the Aptima Combo 2 nucleic acid amplification test in detection of Neisseria gonorrhoeae from genital and extra-genital sites: a retrospective study. Sex Transm Infect. 2012 Feb;88(1):27-31. doi: 10.1136/sextrans-2011-050075. Epub 2011 Oct 27. PMID 22034496
- [Background] Pope CF, Hay P, Alexander S, Capaldi K, Dave J, Sadiq ST, Ison CA, Planche T. Positive predictive value of the Becton Dickinson VIPER system and the ProbeTec GC Q x assay, in extracted mode, for detection of Neisseria gonorrhoeae. Sex Transm Infect. 2010 Nov;86(6):465-9. doi: 10.1136/sti.2010.044065. PMID 20940160
- [Background] Goldenberg SD, Finn J, Sedudzi E, White JA, Tong CY. Performance of the GeneXpert CT/NG assay compared to that of the Aptima AC2 assay for detection of rectal Chlamydia trachomatis and Neisseria gonorrhoeae by use of residual Aptima Samples. J Clin Microbiol. 2012 Dec;50(12):3867-9. doi: 10.1128/JCM.01930-12. Epub 2012 Sep 19. PMID 22993183
- [Background] Boyadzhyan B, Yashina T, Yatabe JH, Patnaik M, Hill CS. Comparison of the APTIMA CT and GC assays with the APTIMA combo 2 assay, the Abbott LCx assay, and direct fluorescent-antibody and culture assays for detection of Chlamydia trachomatis and Neisseria gonorrhoeae. J Clin Microbiol. 2004 Jul;42(7):3089-93. doi: 10.1128/JCM.42.7.3089-3093.2004. PMID 15243065
- [Background] Chernesky MA, Martin DH, Hook EW, Willis D, Jordan J, Wang S, Lane JR, Fuller D, Schachter J. Ability of new APTIMA CT and APTIMA GC assays to detect Chlamydia trachomatis and Neisseria gonorrhoeae in male urine and urethral swabs. J Clin Microbiol. 2005 Jan;43(1):127-31. doi: 10.1128/JCM.43.1.127-131.2005. PMID 15634960
- [Background] Moncada J, Donegan E, Schachter J. Evaluation of CDC-recommended approaches for confirmatory testing of positive Neisseria gonorrhoeae nucleic acid amplification test results. J Clin Microbiol. 2008 May;46(5):1614-9. doi: 10.1128/JCM.02301-07. Epub 2008 Mar 5. PMID 18322062
- [Background] Tabrizi SN, Unemo M, Limnios AE, Hogan TR, Hjelmevoll SO, Garland SM, Tapsall J. Evaluation of six commercial nucleic acid amplification tests for detection of Neisseria gonorrhoeae and other Neisseria species. J Clin Microbiol. 2011 Oct;49(10):3610-5. doi: 10.1128/JCM.01217-11. Epub 2011 Aug 3. PMID 21813721
- [Derived] Doernberg SB, Komarow L, Tran TTT, Sund Z, Pandori MW, Jensen D, Tsalik EL, Deal CD, Chambers HF, Fowler VG, Evans SR, Patel R, Klausner JD. Simultaneous Evaluation of Diagnostic Assays for Pharyngeal and Rectal Neisseria gonorrhoeae and Chlamydia trachomatis Using a Master Protocol. Clin Infect Dis. 2020 Dec 3;71(9):2314-2322. doi: 10.1093/cid/ciz1105. PMID 31734695

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 2767
Completed | 2598
Not Completed | 169

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Arm/Group | Intervention
Number analyzed (Participants) | 2598
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25
  Between 18 and 65 years | 2542
  >=65 years | 31
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [25 to 41]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Man | 2010
  Gender: Woman | 532
  Gender: Transman | 3
  Gender: Transwoman | 42
  Gender: Genderqueer | 8
  Gender: Decline to answer | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 539
  Male | 2059
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 772
  Not Hispanic or Latino | 1814
  Unknown or Not Reported | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 15
  Asian | 84
  Native Hawaiian or Other Pacific Islander | 4
  Black or African American | 935
  White | 1285
  More than one race | 71
  Unknown or Not Reported | 204
Region of Enrollment [Number; unit: participants]
  United States | 2598

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Nucleic Acid Amplification Test (NAAT) 1 Index Test Results Relative to Anatomic Site Infection Status (ASIS) Reference Results for Neisseria Gonorrhoeae (NG) in Pharynx
Description: NAAT 1 index test results include negative, positive, and no result. ASIS reference results are the combination of the NAAT 2 and NAAT 3 index test results. ASIS reference results include negative, positive, indeterminate, and invalid.
Time Frame: One day
Population: Of the 2598 participants who completed the overall study per the Participant Flow module, 8 participants had incomplete test results and were excluded from this outcome.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Performance of nucleic acid amplification test 1 to detect Neisseria gonorrhoeae from swabs collected from the pharynx.
Arm/Group | Intervention
Number analyzed (Participants) | 2590
Participants
  Index Test Negative; ASIS Negative | 2340
  Index Test Negative; ASIS Positive | 9
  Index Test Negative; ASIS Indeterminate | 2
  Index Test Negative; ASIS Invalid | 1
  Index Test Positive; ASIS Negative | 28
  Index Test Positive; ASIS Positive | 195
  Index Test Positive; ASIS Indeterminate | 1
  Index Test Positive; ASIS Invalid | 1
  Index Test No Result; ASIS Negative | 11
  Index Test No Result; ASIS Positive | 0
  Index Test No Result; ASIS Indeterminate | 0
  Index Test No Result; ASIS Invalid | 2
Statistical Analysis 1: Comparison: Intervention; Test type: Other — Estimated positive percent agreement (PPA) defined as: (Index Test Positive; ASIS Positive) / (Index Test Negative; ASIS Positive + Index Test Positive; ASIS Positive + Index Test Negative; ASIS Indeterminate); PPA = 94.7, 95% CI 2-sided [90.7 to 97.0] — PPA estimated with two-sided 95% score confidence interval
Statistical Analysis 2: Comparison: Intervention; Test type: Other — Estimated negative percent agreement (NPA) defined as: (Index Test Negative; ASIS Negative) / (Index Test Negative; ASIS Negative + Index Test Positive; ASIS Negative + Index Test Positive; ASIS Indeterminate); NPA = 98.8, 95% CI 2-sided [98.2 to 99.1] — NPA estimated with two-sided 95% score confidence interval

2. Primary Outcome: Number of Participants With Nucleic Acid Amplification Test (NAAT) 1 Index Test Results Relative to Anatomic Site Infection Status (ASIS) Reference Results for Neisseria Gonorrhoeae (NG) in Rectum
Description: as for outcome 1
Time Frame: One day
Population: Of the 2598 participants who completed the overall study per the Participant Flow module, 13 participants had incomplete test results and were excluded from this outcome.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Performance of nucleic acid amplification test 1 to detect Neisseria gonorrhoeae from swabs collected from the rectum.
Arm/Group | Intervention
Number analyzed (Participants) | 2585
Participants
  Index Test Negative; ASIS Negative | 2323
  Index Test Negative; ASIS Positive | 17
  Index Test Negative; ASIS Indeterminate | 1
  Index Test Negative; ASIS Invalid | 2
  Index Test Positive; ASIS Negative | 8
  Index Test Positive; ASIS Positive | 187
  Index Test Positive; ASIS Indeterminate | 1
  Index Test Positive; ASIS Invalid | 0
  Index Test No Result; ASIS Negative | 40
  Index Test No Result; ASIS Positive | 1
  Index Test No Result; ASIS Indeterminate | 0
  Index Test No Result; ASIS Invalid | 5
Statistical Analysis 1: Comparison: Intervention; Test type: Other — [test comment as in outcome 1, analysis 1]; PPA = 91.2, 95% CI 2-sided [86.5 to 94.4] — PPA estimated with two-sided 95% score confidence interval
Statistical Analysis 2: Comparison: Intervention; Test type: Other — [test comment as in outcome 1, analysis 2]; NPA = 99.6, 95% CI 2-sided [99.3 to 99.8] — NPA estimated with two-sided 95% score confidence interval

3. Primary Outcome: Number of Participants With Nucleic Acid Amplification Test (NAAT) 2 Index Test Results Relative to Anatomic Site Infection Status (ASIS) Reference Results for Neisseria Gonorrhoeae (NG) in Pharynx
Description: NAAT 2 index test results include negative, positive, equivocal, and no result. ASIS reference results are the combination of the NAAT 1 and NAAT 3 index test results. ASIS reference results include negative, positive, indeterminate, and invalid
Time Frame: One day
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Performance of nucleic acid amplification test 2 to detect Neisseria gonorrhoeae from swabs collected from the pharynx.
Arm/Group | Intervention
Number analyzed (Participants) | 2590
Participants
  Index Test Negative; ASIS Negative | 2351
  Index Test Negative; ASIS Positive | 8
  Index Test Negative; ASIS Indeterminate | 2
  Index Test Negative; ASIS Invalid | 2
  Index Test Positive; ASIS Negative | 25
  Index Test Positive; ASIS Positive | 195
  Index Test Positive; ASIS Indeterminate | 1
  Index Test Positive; ASIS Invalid | 0
  Index Test Equivocal; ASIS Negative | 3
  Index Test Equivocal; ASIS Positive | 0
  Index Test Equivocal; ASIS Indeterminate | 0
  Index Test Equivocal; ASIS Invalid | 0
  Index Test No Result; ASIS Negative | 0
  Index Test No Result; ASIS Positive | 1
  Index Test No Result; ASIS Indeterminate | 0
  Index Test No Result; ASIS Invalid | 2
Statistical Analysis 1: Comparison: Intervention; Test type: Other — Estimated positive percent agreement (PPA) defined as: (Index Test Positive; ASIS Positive) / (Index Test Negative; ASIS Positive + Index Test Positive; ASIS Positive + Index Test Equivocal; ASIS Indeterminate + Index Test Negative; ASIS Indeterminate); PPA = 95.1, 95% CI 2-sided [91.3 to 97.3] — PPA estimated with two-sided 95% score confidence interval
Statistical Analysis 2: Comparison: Intervention; Test type: Other — Estimated negative percent agreement (NPA) defined as: (Index Test Negative; ASIS Negative) / (Index Test Negative; ASIS Negative + Index Test Positive; ASIS Negative + Index Test Equivocal; ASIS Negative + Index Test Positive; ASIS Indeterminate); NPA = 98.8, 95% CI 2-sided [98.3 to 99.2] — NPA estimated with two-sided 95% score confidence interval

4. Primary Outcome: Number of Participants With Nucleic Acid Amplification Test (NAAT) 2 Index Test Results Relative to Anatomic Site Infection Status (ASIS) Reference Results for Neisseria Gonorrhoeae (NG) in Rectum
Description: as for outcome 3
Time Frame: One day
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Performance of nucleic acid amplification test 2 to detect Neisseria gonorrhoeae from swabs collected from the rectum.
Arm/Group | Intervention
Number analyzed (Participants) | 2585
Participants
  Index Test Negative; ASIS Negative | 2359
  Index Test Negative; ASIS Positive | 5
  Index Test Negative; ASIS Indeterminate | 0
  Index Test Negative; ASIS Invalid | 3
  Index Test Positive; ASIS Negative | 13
  Index Test Positive; ASIS Positive | 192
  Index Test Positive; ASIS Indeterminate | 2
  Index Test Positive; ASIS Invalid | 0
  Index Test Equivocal; ASIS Negative | 3
  Index Test Equivocal; ASIS Positive | 2
  Index Test Equivocal; ASIS Indeterminate | 0
  Index Test Equivocal; ASIS Invalid | 0
  Index Test No Result; ASIS Negative | 1
  Index Test No Result; ASIS Positive | 0
  Index Test No Result; ASIS Indeterminate | 0
  Index Test No Result; ASIS Invalid | 5
Statistical Analysis 1: Comparison: Intervention; Test type: Other — [test comment as in outcome 1, analysis 1]; PPA = 96.5, 95% CI 2-sided [92.9 to 98.3] — PPA estimated with two-sided 95% score confidence interval
Statistical Analysis 2: Comparison: Intervention; Test type: Other — [test comment as in outcome 1, analysis 2]; NPA = 99.2, 95% CI 2-sided [98.8 to 99.5] — NPA estimated with two-sided 95% score confidence interval

5. Primary Outcome: Number of Participants With Nucleic Acid Amplification Test (NAAT) 3 Index Test Results Relative to Anatomic Site Infection Status (ASIS) Reference Results for Neisseria Gonorrhoeae (NG) in Pharynx
Description: NAAT 3 index test results include negative, positive, and no result. ASIS reference results are the combination of the NAAT 1 and NAAT 2 index test results. ASIS reference results include negative, positive, indeterminate, and invalid.
Time Frame: One day
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Performance of nucleic acid amplification test 3 to detect Neisseria gonorrhoeae from swabs collected from the pharynx.
Arm/Group | Intervention
Number analyzed (Participants) | 2590
Participants
  Index Test Negative; ASIS Negative | 2356
  Index Test Negative; ASIS Positive | 28
  Index Test Negative; ASIS Indeterminate | 4
  Index Test Negative; ASIS Invalid | 1
  Index Test Positive; ASIS Negative | 11
  Index Test Positive; ASIS Positive | 179
  Index Test Positive; ASIS Indeterminate | 0
  Index Test Positive; ASIS Invalid | 1
  Index Test No Result; ASIS Negative | 6
  Index Test No Result; ASIS Positive | 2
  Index Test No Result; ASIS Indeterminate | 0
  Index Test No Result; ASIS Invalid | 2
Statistical Analysis 1: Comparison: Intervention; Test type: Other — [test comment as in outcome 1, analysis 1]; PPA = 84.8, 95% CI 2-sided [79.4 to 89.0] — PPA estimated with two-sided 95% score confidence interval
Statistical Analysis 2: Comparison: Intervention; Test type: Other — [test comment as in outcome 1, analysis 2]; NPA = 99.5, 95% CI 2-sided [99.2 to 99.7] — NPA estimated with two-sided 95% score confidence interval

6. Primary Outcome: Number of Participants With Nucleic Acid Amplification Test (NAAT) 3 Index Test Results Relative to Anatomic Site Infection Status (ASIS) Reference Results for Neisseria Gonorrhoeae (NG) in Rectum
Description: as for outcome 5
Time Frame: One day
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Performance of nucleic acid amplification test 3 to detect Neisseria gonorrhoeae from swabs collected from the rectum.
Arm/Group | Intervention
Number analyzed (Participants) | 2585
Participants
  Index Test Negative; ASIS Negative | 2312
  Index Test Negative; ASIS Positive | 23
  Index Test Negative; ASIS Indeterminate | 1
  Index Test Negative; ASIS Invalid | 1
  Index Test Positive; ASIS Negative | 8
  Index Test Positive; ASIS Positive | 181
  Index Test Positive; ASIS Indeterminate | 2
  Index Test Positive; ASIS Invalid | 0
  Index Test No Result; ASIS Negative | 51
  Index Test No Result; ASIS Positive | 1
  Index Test No Result; ASIS Indeterminate | 0
  Index Test No Result; ASIS Invalid | 5
Statistical Analysis 1: Comparison: Intervention; Test type: Other — [test comment as in outcome 1, analysis 1]; PPA = 88.3, 95% CI 2-sided [83.2 to 92.0] — PPA estimated with two-sided 95% score confidence interval
Statistical Analysis 2: Comparison: Intervention; Test type: Other — [test comment as in outcome 1, analysis 2]; NPA = 99.6, 95% CI 2-sided [99.2 to 99.8] — NPA estimated with two-sided 95% score confidence interval

7. Primary Outcome: Number of Participants With Nucleic Acid Amplification Test (NAAT) 1 Index Test Results Relative to Anatomic Site Infection Status (ASIS) Reference Results for Chlamydia Trachomatis (CT) in Pharynx
Description: as for outcome 1
Time Frame: One day
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Performance of nucleic acid amplification test 1 to detect Chlamydia trachomatis from swabs collected from the pharynx.
Arm/Group | Intervention
Number analyzed (Participants) | 2590
Participants
  Index Test Negative; ASIS Negative | 2518
  Index Test Negative; ASIS Positive | 2
  Index Test Negative; ASIS Indeterminate | 0
  Index Test Negative; ASIS Invalid | 2
  Index Test Positive; ASIS Negative | 6
  Index Test Positive; ASIS Positive | 47
  Index Test Positive; ASIS Indeterminate | 2
  Index Test Positive; ASIS Invalid | 0
  Index Test No Result; ASIS Negative | 11
  Index Test No Result; ASIS Positive | 0
  Index Test No Result; ASIS Indeterminate | 0
  Index Test No Result; ASIS Invalid | 2
Statistical Analysis 1: Comparison: Intervention; Test type: Other — [test comment as in outcome 1, analysis 1]; PPA = 95.9, 95% CI 2-sided [86.3 to 98.9] — PPA estimated with two-sided 95% score confidence interval
Statistical Analysis 2: Comparison: Intervention; Test type: Other — [test comment as in outcome 1, analysis 2]; NPA = 99.7, 95% CI 2-sided [99.4 to 99.8] — NPA estimated with two-sided 95% score confidence interval

8. Primary Outcome: Number of Participants With Nucleic Acid Amplification Test (NAAT) 1 Index Test Results Relative to Anatomic Site Infection Status (ASIS) Reference Results for Chlamydia Trachomatis (CT) in Rectum
Description: as for outcome 1
Time Frame: One day
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Performance of nucleic acid amplification test 1 to detect Chlamydia trachomatis from swabs collected from the rectum.
Arm/Group | Intervention
Number analyzed (Participants) | 2585
Participants
  Index Test Negative; ASIS Negative | 2292
  Index Test Negative; ASIS Positive | 28
  Index Test Negative; ASIS Indeterminate | 4
  Index Test Negative; ASIS Invalid | 2
  Index Test Positive; ASIS Negative | 15
  Index Test Positive; ASIS Positive | 197
  Index Test Positive; ASIS Indeterminate | 1
  Index Test Positive; ASIS Invalid | 0
  Index Test No Result; ASIS Negative | 40
  Index Test No Result; ASIS Positive | 1
  Index Test No Result; ASIS Indeterminate | 0
  Index Test No Result; ASIS Invalid | 5
Statistical Analysis 1: Comparison: Intervention; Test type: Other — [test comment as in outcome 1, analysis 1]; PPA = 86.0, 95% CI 2-sided [80.9 to 89.9] — PPA estimated with two-sided 95% score confidence interval
Statistical Analysis 2: Comparison: Intervention; Test type: Other — [test comment as in outcome 1, analysis 2]; NPA = 99.3, 95% CI 2-sided [98.9 to 99.6] — NPA estimated with two-sided 95% score confidence interval

9. Primary Outcome: Number of Participants With Nucleic Acid Amplification Test (NAAT) 2 Index Test Results Relative to Anatomic Site Infection Status (ASIS) Reference Results for Chlamydia Trachomatis (CT) in Pharynx
Description: as for outcome 3
Time Frame: One day
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Performance of nucleic acid amplification test 2 to detect Chlamydia trachomatis from swabs collected from the pharynx.
Arm/Group | Intervention
Number analyzed (Participants) | 2590
Participants
  Index Test Negative; ASIS Negative | 2526
  Index Test Negative; ASIS Positive | 6
  Index Test Negative; ASIS Indeterminate | 0
  Index Test Negative; ASIS Invalid | 2
  Index Test Positive; ASIS Negative | 8
  Index Test Positive; ASIS Positive | 45
  Index Test Positive; ASIS Indeterminate | 0
  Index Test Positive; ASIS Invalid | 0
  Index Test Equivocal; ASIS Negative | 0
  Index Test Equivocal; ASIS Positive | 0
  Index Test Equivocal; ASIS Indeterminate | 0
  Index Test Equivocal; ASIS Invalid | 0
  Index Test No Result; ASIS Negative | 1
  Index Test No Result; ASIS Positive | 0
  Index Test No Result; ASIS Indeterminate | 0
  Index Test No Result; ASIS Invalid | 2
Statistical Analysis 1: Comparison: Intervention; Test type: Other — [test comment as in outcome 3, analysis 1]; PPA = 88.2, 95% CI 2-sided [76.6 to 94.5] — PPA estimated with two-sided 95% score confidence interval
Statistical Analysis 2: Comparison: Intervention; Test type: Other — [test comment as in outcome 3, analysis 2]; NPA = 99.7, 95% CI 2-sided [99.4 to 99.8] — NPA estimated with two-sided 95% score confidence interval

10. Primary Outcome: Number of Participants With Nucleic Acid Amplification Test (NAAT) 2 Index Test Results Relative to Anatomic Site Infection Status (ASIS) Reference Results for Chlamydia Trachomatis (CT) in Rectum
Description: as for outcome 3
Time Frame: One day
Population: Of the 2598 participants who completed the overall study per the Participant Flow module, 13 participants had incomplete test results and were excluded from analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Performance of nucleic acid amplification test 2 to detect Chlamydia trachomatis from swabs collected from the rectum.
Arm/Group | Intervention
Number analyzed (Participants) | 2585
Participants
  Index Test Negative; ASIS Negative | 2322
  Index Test Negative; ASIS Positive | 18
  Index Test Negative; ASIS Indeterminate | 2
  Index Test Negative; ASIS Invalid | 3
  Index Test Positive; ASIS Negative | 25
  Index Test Positive; ASIS Positive | 197
  Index Test Positive; ASIS Indeterminate | 0
  Index Test Positive; ASIS Invalid | 0
  Index Test Equivocal; ASIS Negative | 5
  Index Test Equivocal; ASIS Positive | 5
  Index Test Equivocal; ASIS Indeterminate | 2
  Index Test Equivocal; ASIS Invalid | 0
  Index Test No Result; ASIS Negative | 1
  Index Test No Result; ASIS Positive | 0
  Index Test No Result; ASIS Indeterminate | 0
  Index Test No Result; ASIS Invalid | 5
Statistical Analysis 1: Comparison: Intervention; Test type: Other — [test comment as in outcome 3, analysis 1]; PPA = 88.7, 95% CI 2-sided [83.9 to 92.3] — PPA estimated with two-sided 95% score confidence interval
Statistical Analysis 2: Comparison: Intervention; Test type: Other — [test comment as in outcome 3, analysis 2]; NPA = 98.7, 95% CI 2-sided [98.2 to 99.1] — NPA estimated with two-sided 95% score confidence interval

11. Primary Outcome: Number of Participants With Nucleic Acid Amplification Test (NAAT) 3 Index Test Results Relative to Anatomic Site Infection Status (ASIS) Reference Results for Chlamydia Trachomatis (CT) in Pharynx
Description: NAAT 3 index test results include negative, positive, equivocal, and no result. ASIS reference results are the combination of the NAAT 1 and NAAT 2 index test results. ASIS reference results include negative, positive, indeterminate, and invalid.
Time Frame: One day
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Performance of nucleic acid amplification test 3 to detect Chlamydia trachomatis from swabs collected from the pharynx.
Arm/Group | Intervention
Number analyzed (Participants) | 2590
Participants
  Index Test Negative; ASIS Negative | 2522
  Index Test Negative; ASIS Positive | 8
  Index Test Negative; ASIS Indeterminate | 0
  Index Test Negative; ASIS Invalid | 2
  Index Test Positive; ASIS Negative | 4
  Index Test Positive; ASIS Positive | 42
  Index Test Positive; ASIS Indeterminate | 1
  Index Test Positive; ASIS Invalid | 0
  Index Test Equivocal; ASIS Negative | 1
  Index Test Equivocal; ASIS Positive | 0
  Index Test Equivocal; ASIS Indeterminate | 0
  Index Test Equivocal; ASIS Invalid | 0
  Index Test No Result; ASIS Negative | 7
  Index Test No Result; ASIS Positive | 1
  Index Test No Result; ASIS Indeterminate | 0
  Index Test No Result; ASIS Invalid | 2
Statistical Analysis 1: Comparison: Intervention; Test type: Other — [test comment as in outcome 3, analysis 1]; PPA = 84.0, 95% CI 2-sided [71.5 to 91.7] — PPA estimated with two-sided 95% score confidence interval
Statistical Analysis 2: Comparison: Intervention; Test type: Other — [test comment as in outcome 3, analysis 2]; NPA = 99.8, 95% CI 2-sided [99.5 to 99.9] — NPA estimated with two-sided 95% score confidence interval

12. Primary Outcome: Number of Participants With Nucleic Acid Amplification Test (NAAT) 3 Index Test Results Relative to Anatomic Site Infection Status (ASIS) Reference Results for Chlamydia Trachomatis (CT) in Rectum
Description: as for outcome 11
Time Frame: One day
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Performance of nucleic acid amplification test 3 to detect Chlamydia trachomatis from swabs collected from the rectum.
Arm/Group | Intervention
Number analyzed (Participants) | 2585
Participants
  Index Test Negative; ASIS Negative | 2277
  Index Test Negative; ASIS Positive | 34
  Index Test Negative; ASIS Indeterminate | 5
  Index Test Negative; ASIS Invalid | 1
  Index Test Positive; ASIS Negative | 19
  Index Test Positive; ASIS Positive | 190
  Index Test Positive; ASIS Indeterminate | 2
  Index Test Positive; ASIS Invalid | 0
  Index Test Equivocal; ASIS Negative | 0
  Index Test Equivocal; ASIS Positive | 0
  Index Test Equivocal; ASIS Indeterminate | 0
  Index Test Equivocal; ASIS Invalid | 0
  Index Test No Result; ASIS Negative | 49
  Index Test No Result; ASIS Positive | 2
  Index Test No Result; ASIS Indeterminate | 1
  Index Test No Result; ASIS Invalid | 5
Statistical Analysis 1: Comparison: Intervention; Test type: Other — [test comment as in outcome 3, analysis 1]; PPA = 83.0, 95% CI 2-sided [77.6 to 87.3] — PPA estimated with two-sided 95% score confidence interval
Statistical Analysis 2: Comparison: Intervention; Test type: Other — [test comment as in outcome 3, analysis 2]; NPA = 99.1, 95% CI 2-sided [98.6 to 99.4] — NPA estimated with two-sided 95% score confidence interval

ADVERSE EVENTS:
Time Frame: One day
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/2598
Serious Adverse Events (participants affected / at risk) | 0/2598
Other Adverse Events (participants affected / at risk) | 0/2598

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following completion of the study, the Investigator may publish the results of this research under the oversight of the Antibiotic Resistance Leadership Group (ARLG) Publication Committee. All public presentations by participating Investigators, participating institutions, SDMC, and ARLG, that use ARLG data and are intended to represent the ARLG, or are supported by the ARLG, will be reviewed by the ARLG Publication Committee per the ARLG Publication Committee Charter.

DOCUMENTS (2):
  • Study Protocol (2017-12-04): https://cdn.clinicaltrials.gov/large-docs/01/NCT02870101/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/01/NCT02870101/SAP_001.pdf